CLINICAL TRIAL: NCT06731348
Title: Patient Satisfaction With Opioid Restriction After Urogynecologic Surgery: A Randomized Non-Inferiority Trial
Brief Title: Patient Satisfaction With Opioid Restriction After Urogynecologic Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2024-0454
Record Dates: First submitted 2024-11-04; First posted 2024-12-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-12

CONDITIONS: Patient Satisfaction; Opioid Use After Surgery; Urogynecologic Surgery
Keywords: Patient Satisfaction; Opioid Use after Urogynecologic Surgery
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Opioid Prescribing - Oxycodone HCl 5mg (Active Comparator): Participants will receive standard opioid prescribing - Oxycodone 5mg x10 tablets for major cases, 5 tablets for minor cases.
  Interventions: Drug: standard opioid prescribing
- Restricted Opioid Prescribing - Oxycodone HCl 5mg (Experimental): Participants in the restricted opioid prescribing group will receive restricted opioid prescribing after surgery. They will receive 1 tablet of Oxycodone HCl 5mg
  Interventions: Drug: restricted opioid prescribing

INTERVENTIONS:
Drug: restricted opioid prescribing — Participants in the restricted opioid prescribing group will receive restricted opioid prescribing after surgery. They will receive 1 tablet of Oxycodone HCl 5mg.
  Arms: Restricted Opioid Prescribing - Oxycodone HCl 5mg
Drug: standard opioid prescribing — Participants will receive standard opioid prescribing - Oxycodone HCl 5mg x10 tablets for major cases, 5 tablets for minor cases.
  Arms: Standard Opioid Prescribing - Oxycodone HCl 5mg

SUMMARY:
Patients undergoing surgery with the Walter Reed National Military Medical Center Urogynecology Clinic will be randomized to either standard opioid prescribing or restricted opioid prescribing. They will be surveyed on their satisfaction with their postoperative pain control and their pain levels and opioid use will be tracked postoperatively.

DETAILED DESCRIPTION:
This study is a 2 arm, unmasked, single center, randomized controlled, non-inferiority study comparing participant satisfaction with post-operative pain control between participants randomized to a restrictive opioid prescribing protocol versus a standard opioid prescribing protocol.

All females aged 18 years and older who are scheduled for a minor or major urogynecologic surgery who are receiving care at Walter Reed National Military Medical Center (WRNMMC) Urogynecology clinic will be eligible for the study. Of note, all those seen in the WRNMMC Urogynecologic clinic are female. Minor surgeries will include colporrhaphy, midurethral sling placement, vaginal mesh removal or revision, urethral diverticulectomy, or vaginal cyst excision. Major surgeries will include vaginal vault suspension, minimally invasive (laparoscopic or robotic) sacrocolpopexy, minimally invasive (laparoscopic or robotic) hysteropexy, and colpocleisis. Major cases may or may not include hysterectomy and/or bilateral salpingectomy at the time of surgery.

Prior to the scheduled surgical procedure, the participant will present for an in-person, routine pre-operative appointment which is standard of care in our practice and involves a review of the participant's histories and medications, as well as signing surgical consents and reviewing pre- and post-operative instructions. All participants will receive standardized pre-operative and post-operative counseling as is standard of care in our clinical practice.

Participants will be randomized to determine the protocol assignment - standard opioid prescribing or restricted opioid prescribing. Standard opioid prescribing participants will be prescribed the standard opioid prescription - 5 tablets of Oxycodone HCl 5mg for minor procedures, 10 tablets of Oxycodone HCl 5mg for major procedures - for post-operative pain control. Restricted opioid prescribing participants will be prescribed 1 tablet of Oxycodone HCl 5mg for both minor and major procedures.

Participants will follow-up at 7-10 days and 6-8 weeks to determine their satisfaction with their post-operative pain control, as well as their pain levels and opioid use post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age and older
* Scheduled for urogynecologic surgical procedure
* Ability to follow study instructions and complete all required follow-up
* DEERS eligible
* Willing to take the SOC opioid dose or the restricted dose

Exclusion Criteria:

* Ineligible for non-opioid pain medication, including allergy to acetaminophen or NSAIDS
* History of opioid abuse determined by asking the potential participant about history of opioid abuse and reviewing potential participant's chart to look for prior or active diagnosis of opioid abuse.
* Females who are breastfeeding, pregnant or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study
* Inability to speak or read English. Non-English speakers will be excluded from this study for ease of being able to allow the principal investigator to communicate with the patients during the consents, initial and all follow-up communication. Some of the questionnaires used have also only been validated in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with post-operative pain control | post-operative day 7-10
  Satisfaction with post-operative pain control on post-operative day (POD) 7-10 in participants undergoing urogynecologic surgery who receive either the routine opioid prescribing protocol or the restrictive prescribing protocol.

SECONDARY OUTCOMES:
Participant satisfaction with post-operative pain control at 6-8 weeks post-operatively | post-operative weeks 6-8
Difference in satisfaction with post-operative pain control between POD 7-10 and 6-8 weeks post-operatively. | post-operative week 6-8
Post-operative opioid use on POD 1-7 | post-operative days 1-7
Patient pain scores on POD 1-7 | post-operative days 1-7
Postoperative opioid refill rates over 6 weeks post-operatively | post-operative week 6
Participant utilization of health care resources over 6 weeks post-operatively. | post-operative week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No